CLINICAL TRIAL: NCT01715636
Title: Safety, Tolerability, and Adherence to Co-formulated Emtricitabine-rilpivirine-tenofovir Used as HIV Nonoccupational Post Exposure Prophylaxis in Men Who Have Sex With Men (EPEP)
Brief Title: Safety, Tolerability,and Adherence to Co-formulated Tenofovir-emtricitabine-rilpivirine Used as HIV Nonoccupational Post-exposure Prophylaxis in Men Who Have Sex With Men.
Acronym: EPEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrew Carr (Other)
Responsible Party: Sponsor-Investigator, Andrew Carr, Professor, St Vincent's Hospital
Organization: St Vincent's Hospital, Sydney (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1.0 dated 28 May 2012; Carr (IN-AU-264-0119) (Other Grant/Funding Number: Gilead Sciences Pty Ltd)
Record Dates: First submitted 2012-10-18; First posted 2012-10-29 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: HIV Nonoccupational Post-exposure Prophylaxis in Men Who Have Sex With Men
MeSH Terms: interventions — Rilpivirine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eviplera (Other): Eviplera = emtricitabine 200mg, rilpivirine 25mg, tenofovir 245mg, one tablet, once daily, taken with food, for 28 days
  Interventions: Drug: Eviplera = emtricitabine 200mg, rilpivirine 25mg, tenofovir 245mg

INTERVENTIONS:
Drug: Eviplera = emtricitabine 200mg, rilpivirine 25mg, tenofovir 245mg
  Other Names: Eviplera

SUMMARY:
This study aims to describe the safety, tolerability and adherence to the coformulated anti-HIV drug tenofovir-emtricitabine-rilpivirine (eviplera) when given to men who have sex with men (MSM) following an actual or potential sexual exposure to HIV. This biomedical intervention is known as nonoccupational post-exposure prophylaxis (NPEP). Patients receive NPEP if they meet the criteria outlined in the 2007 National Australian NPEP Guidelines. Three or two anti-HIV drugs are administered for 28-days depending on the severity of the the assessed HIV acquisition risk. In this study eviplera would constitute 3-drug NPEP. Tenofovir-emtricitabine (truvada) a component of eviplera has been used in NPEP at SVH since 2006.

This is a multi site, prospective, open-label, non-randomised trial. Participants will be MSM who present at the various recruitment sites requesting NPEP. Initially, 50 eligible participants will be assigned to receive eviplera 25mg once daily taken with food for 28-days according to established Australian guidelines for the use of 3-drug NPEP. There will be 7 visits over a 12-week period. Follow-up post NPEP is for 8 weeks. If an interim analysis demonstrates acceptable safety, it is proposed to seek ethics approval to increase the samples size to 100 patients to gain more accurate information on regimen completion rate and on-drug adherence.

The primary study objectives are:

1. To describe the safety of 28 days of NPEP using co-formulated FTC-RPV-TDF
2. To describe the tolerability of 28 days of NPEP using FTC-RPV-TDF
3. To describe on-drug adherence and regimen completion rates of 28 days of NPEP using FTC-RPV-TDF

ELIGIBILITY:
Inclusion Criteria:

1. Man who has sex with men
2. Age at least 18 years
3. Eligible for 3-drug NPEP according to Australian guidelines for the use of 3-drug NPEP following an actual or potential sexual exposure to HIV or receptive anal intercourse with an unknown source
4. Able to provide written, informed consent
5. Able to commit to the study visits

   Exclusion Criteria:
6. Non-sexual exposure
7. Exposure occurring during sex between a man and a woman
8. HIV infection diagnosed on day 1 serological testing including indeterminate serology consistent with possible primary HIV infection
9. Use of any medication contraindicated with FTC-RPV-TDF
10. Serum hepatic transaminase (alanine aminotransferase [ALT] greater than 5 times the upper limit of the normal range
11. Serum estimated Glomerular Filtration Rate (eGFR) <60mL/min/ BSAc
12. Current therapy for hepatitis B
13. Day 1 serological evidence of chronic/active hepatitis B
14. Previous NPEP containing FTC-RPV-TDF
15. A patient with a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To describe the safety of 28 days of nonoccupational post-exposure prophylaxis with Eviplera | 28 days
  Objective AE and SAE data collection/grading utilising DAIDS data collection tool. Measurement of weight, electrolytes, urea, creatinine, eGFR, inorganic phosphate, calcium, liver function, glucose, amylase, lipase, creatine kinase, lactate

SECONDARY OUTCOMES:
To describe the tolerability of 28 days of nonoccupational post-exposure prophylaxis with Eviplera | 28 days
  Subjective reporting of AEs with data collection/grading utilising DAIDS-AE

OTHER OUTCOMES:
on-drug adherence and regimen completion dates | 28 days

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Sydney Sexual Heatlh Centre, Sydney, New South Wales
  - St Vincents Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Melbourne Sexual Health Centre, Melbourne, Victoria

REFERENCES:
- [Derived] Foster R, McAllister J, Read TR, Pierce AB, Richardson R, McNulty A, Carr A. Single-Tablet Emtricitabine-Rilpivirine-Tenofovir as HIV Postexposure Prophylaxis in Men Who Have Sex With Men. Clin Infect Dis. 2015 Oct 15;61(8):1336-41. doi: 10.1093/cid/civ511. Epub 2015 Jun 29. PMID 26123937